CLINICAL TRIAL: NCT00670891
Title: A Prospective, Non-Randomized, Open-Label Study on the Clinical Effects of Hyperbaric Oxygen Therapy in Thai Autistic Children
Brief Title: A Clinical Trial of the Clinical Effects of Hyperbaric Oxygen Therapy in Thai Autistic Children
Acronym: VPH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vachira Phuket Hospital (Other)
Responsible Party: HBOT and Developmental Clinic Team, Vachira Phuket Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VP 000001
Record Dates: First submitted 2008-04-29; First posted 2008-05-02 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-04

CONDITIONS: Autistic Disorder
MeSH Terms: conditions — Autistic Disorder | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HBOT (Experimental): HBOT
  Interventions: Procedure: oxygen (Hyperbaric Oxygen Therapy)

INTERVENTIONS:
Procedure: oxygen (Hyperbaric Oxygen Therapy) — Current Accepted Applications of HBOT (2008) Jan 2003, ANDI International
  1. Air or Gas Embolus
  2. Decompression Illness
  3. Carbon Monoxide poising
  4. Clostridial Myonecrosis (Gas Gangrene)
  5. Necrotizing Fasciitis
  6. Crush Injury (Compartment syndromes)
  7. Selected Problem Wounds
  8. Compromised Skin Flaps or Grafts
  9. Refractory Osteomyelitis
  10. Exceptional Anemia due to Blood loss
  11. Osteoradionecrosis
  12. Thermal Burns and Radiation Tissue Damage
  13. Diabetic Wounds
  14. Intra-Cranial Abscess
  15. Brain Injury and other Head Trauma
  16. Cerebral Palsy
  17. High Altitude Sickness
  18. Lyme disease
  Other Names: HBOT

SUMMARY:
Autism is a developmental and behavioral pattern which includes the triad of impairments, 1. social interaction 2. social communication 3. imagination. Inevitable difficulties in the treatment, managing and handle with autistic children are the main problems. Their memories are seemingly in picture or photo records, which are difference from normal population. There are many concepts but no concise in causative factors, including useful treatments, useless and prolong remaining in many studies.

HBOT (Hyperbaric Oxygen Therapy) is a quite modern treatment in Thailand for nitrogen imbalance (decompression sickness syndrome or Caisson disease). How can we apply it to treat the autism? A hypothesis shows evidence that neurons surrounding the permanently damaged epicenter of injury can be reactivated with increased oxygen. Oxygen exists in the blood in two forms, combined with hemoglobin and dissolved in plasma. More oxygen is transported by hemoglobin, but oxygen is delivered to the tissues in dissolved form by the liquid portion of blood. HBOT can increase in plasma oxygen to the tissues including the brain. A little change in oxygen can make the better improvements in : cognitive ability, socialization, sleep, calmness, decreased stimming and language. It can make increased in Glutathione (GSH), and Glutathione (GSH) can decreased in oxidative stress with effected to remove metal compounds (mercury) to improve the autism.

This clinical trial study divided into 3 group populations 1. general autism 2. post-treatment chiropractic autism 3. medicated autism. This comparative study shows the major clinical symptoms before and after the treatment with HBOT. This study results and analysis are the most important for our further projects planning.

DETAILED DESCRIPTION:
Detailed Description There is a general agreement that early identification of autistic spectrum disorders in children and intervention is extremely important.

We would like to find out beneficial effects for early identification and treatment in the autism. Another meaning, it declares that the autism is treatable and can be prevention in the early stage of the symptoms. According to many studies, they had shown brain injury could be caused by heavy metal effects, chemical poisoning, infection, autoimmune response, poor blood flow, lack of oxygen. There are many alternative therapies that were claimed to have some effects to make better results in autistic symptoms, but no definite one which could absolutely cured to the autism.

HBOT (Hyperbaric Oxygen Therapy) is a new way in the treatment for decompression sickness syndrome (Caisson disease) and it can be applied to intervene or concomitant treatments with some symptoms such as diabetic wounds, burnt wounds.

Vachira Phuket Hospital, HBOT center and child development center was established in 2002. This HBOT center is the only one stand-alone center of provincial hospitals in Thailand. Enthusiastic questions in our proceedings were how to declare our opportunities to be a center in HBOT and child developmental center.

If HBOT can be an effective method in alternative therapies, we can help our numerous autistic children. In our proceeding study we found that HBOT was the least interesting method of alternative therapies for the autism in parental opinions. (Figure 1.)

1. General information, the most of sampling groups (75.68%) are female, 40.54% of aged-groups are 30-40 years old, 37.84% of occupations are employee and 32.43% of educations are primary school.
2. Information about opinion of alternative therapies, the most of parents think that the music therapy is the best way. The second is Chiropractic and the third is Art therapy but Animal therapy with the pony is the least effective way.

In the topic of the knowledge about Alternative therapies, the most of parents know about Chiropractic, Art therapy and Music therapy as sequence. The parents know Hyperbaric Oxygen Therapy as the least.

They interested in Music therapy, Chiropractic and Art therapy as sequence. But they are interested in animal therapy with pony and dog as the least. The researchers think that the parents' knowledge about each therapy affects their decision making to choose for their children. Vachira Phuket Hospital has Hyperbaric oxygen therapy (Chamber) which is the new therapy for Autistic children but the parents don't have the knowledge about it. So, the researchers wonder how should we give the information to the parents in order to get the most benefit from this therapy.

Figure 1. Autistic parental attitude surveys in effective, knowledge and interesting in various therapies at Vachira Phuket Hospital, July 2007

Whatever it is our opportunities to prove how effective of HBOT in the treatment for autism and represent autistic pathology mechanisms in preceding hypotheses.

Advantages

1. Administrator's support is provided.
2. Equipment (HBOT) is in the same place with Development Training Clinic.
3. Study by professional physicians in various associated experiences and the developmental nurse, psychologist who accustom with children and the parents (caretakers).
4. Convenience in transportation, which is in a small province.
5. This HBOT is solitary equipment, governed beneath Thailand Ministry of Public Health.

Disadvantages

1. Publication in knowledge about HBOT is very low in Thailand.
2. Harmful may be unknown hidden.
3. Stigmatization is a delicate point in the parents of these children.
4. Worrying and guilty feelings are easily occurred in the parents when something may be unexpected happening.
5. A small province liked Phuket may be difficult to find volunteers for research or study's enrollment.
6. Information gathering and assessment processes including scoring forms may be underneath standardization and not up-to-date.

Problems-solving plans

1. Informed knowledge about HBOT, more and more, to the parents and community.
2. Pre-treatment evaluation was carefully evaluated according to good clinical practice.
3. Respected to their honour, patient's right and kept confidential of the volunteers.
4. Reassured the parents and clarified in details of their concerned issues. Explained the strategies explicitly and slowly.
5. Therefore studied in a small group, closed observation was applied to integrated in details for descriptive study in the volunteers.
6. It could be a pilot study if their any parts of this study were not clearly understood. And thereafter, study planning in the future will be done in the advance conforming design and methodology following our knowledgeable experiences.

ELIGIBILITY:
Inclusion criteria:

1. Both sexes
2. All aged-group
3. All educated group
4. Diagnosis - Autistic disorder, Autistic spectrums
5. Major symptoms - delayed development, delayed speech

Exclusion criteria:

1. Uncontrolled severe explosive behaviours
2. Uncontrolled organic or physical symptoms such as seizure, ear infection
3. Severe phobic or fearful symptoms
4. No parent or caretaker

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2007-07; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Developmental and Skill training assessment, Rajanukul Hospital 5th edition | 10 sessions assessment

SECONDARY OUTCOMES:
Developmental and Skill training assessment, Rajanukul Hospital 5th edition | 20 sessions assessment

CONTACTS AND LOCATIONS:
Overall Officials: Jessada Chungpaibulpatana, MD., Principal Investigator — Vachira Phuket Hospital
Locations (1):
- Vachira Phuket Hospital, Phuket, Phuket, Thailand